CLINICAL TRIAL: NCT04853173
Title: Modality of Pain Management in Ambulatory Tonsillectomy Surgery in Adults: External Pilot Study
Brief Title: Modality of Pain Management in Ambulatory Tonsillectomy Surgery in Adults
Acronym: DACAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/542
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Tonsillar Disorder

STUDY DESIGN:
Intervention Model Description: Assess pain management modalities in adult outpatient tonsillectomy surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ambulatory protocol after adult tonsillectomy (Experimental): prescription of analgesics for outpatient procedure with hospital surveillance
  Interventions: Other: Assess pain management modalities in adult outpatient tonsillectomy surgery

INTERVENTIONS:
Other: Assess pain management modalities in adult outpatient tonsillectomy surgery — use a post-operative analgesia protocol suitable for outpatient surgery. Namely a protocol of analgesia based on the taking of drugs per bone (by mouth) and not intravenous. Pain evaluation.

SUMMARY:
No SFORL recommendation for adult ambulatory tonsillectomy. This study would allow the establishment of an ambulatory management during an adult tonsillectomy. This would allow a return home from J0 for the patient and therefore would improve the comfort of the patients and reduce the cost associated with a conventional hospitalization over several days.

ELIGIBILITY:
Inclusion Criteria:

* programmed Tonsillectomy surgery

Exclusion Criteria:

* Congenital or acquired hemostasis disorder
* Indication of uvulo-bike-pharyngo-plasty
* Contraindication to the use of one of the protocol molecules including pregnancy
* Allergy to analgesic treatments used in the study
* Ongoing analgesic treatment that cannot be interrupted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess pain management modalities in ambulatory tonsillectomy surgery in adults through post-operative pain assessment, with a defined analgesia and anesthesia protocol adapted to ambulatory management. | 14 days
  Pain measured by self-assessment by Analog Visual Scale (0-10). If score is under 4 = efficacity of ansthesia protocol

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No